CLINICAL TRIAL: NCT05772273
Title: Efficacy and Safety of PD-1 Inhibitor, Azacitidine and Low-dose DLI in AML Relapse After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: PD-1 Inhibitor, Azacitidine and Low-dose DLI in AML Relapse After Allo-HSCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-AML-Ⅱ-002
Record Dates: First submitted 2023-02-27; First posted 2023-03-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: PD-1 inhibitor; Azacitidine; low-dose DLI
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Azacitidine and low-dose Donor lymphocyte infusion (Experimental): Patients are given azacytidine for 7 days, followed by 4 DLI treatments on Days 10, 17, 24 and 31, with the dose of DLI and Camrelizumab adjusted according to the donor source. Camrelizumab infusions were given 3 hours after completion of the 1st and 3rd DLIs, respectively.
  Interventions: Drug: Azacitidine; Biological: Donor lymphocyte infusion; Drug: Camrelizumab

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 75 mg/m2 subcutaneously once daily on days 1-7.
Biological: Donor lymphocyte infusion — The 4 DLI doses (dose range: ±10%) of sib-matched donor HSCT patients were 1×10^6/kg, 5×10^6/kg, 1×10^7/kg, 5×10^7/kg; The 4 DLI doses (dose range: ±10%) of haploidentical or unrelated donor HSCT patients were 1×10^5/kg, 5×10^5/kg, 1×10^6/kg, 5×10^6/kg.
Drug: Camrelizumab — Camrelizumab 200mg Q2W for sib-matched donor HSCT patients, 100mg Q2W for haploidentical or unrelated donor HSCT patients.

SUMMARY:
This study aims to evaluate the efficacy and safety of PD-1 inhibitor, Azacitidine, and low-dose DLI in AML relapse After allogeneic hematopoietic stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of AML relapse after allogeneic hematopoietic stem cell transplantation.
2. Adequate organ function.
3. Be able to understand and sign informed consent.
4. Age 18 to 60 years old.
5. Serum pregnancy test for females of childbearing potential that is negative within one week prior to initiation of first dose of treatment. Female patients of childbearing potential and sexually active males must agree to use a highly effective method of contraception throughout the study and for at least 90 days after the last dose of assigned treatment.
6. ECOG performance status ≤ 1.
7. Known HLA-matched donor without contraindications to donate.
8. Life expectancy > 3 months.

Exclusion Criteria:

1. Diagnosis of anther malignant disease.
2. Suspected or proven acute or chronic GVHD.
3. Proven central nervous system leukemia.
4. Prior treatment with anti-PD-1, anti-PD-L1, or DLI.
5. HLA loss positive.
6. Known active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B (HBV) or C (HCV) or Corona Virus Disease 2019(COVID-19);
7. Uncontrolled systemic fungal, bacterial, or viral infection.
8. Known or suspected hypersensitivity to PD-1 inhibitor or azacytidine.
9. Participation in another clinical study within 3 months.
10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | ORR assessment is at day 39 (±2).
  The overall response (completed remission, completed remission with incomplete blood count recovery)

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  OS is measured from the time of enrollment to this trial to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
Progression-Free Survival (PFS) | 2 years
  PFS is measured from the time of enrollment to this study to progression or death.
Adverse events | 1 month
  It is evaluated and graded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China